CLINICAL TRIAL: NCT00212121
Title: Radiation Dose Intensity Study in Breast Cancer in Young Women: a Randomized Phase III Trial of Additional Dose to the Tumor Bed
Brief Title: Radiation Dose Intensity Study in Breast Cancer in Young Women
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M03RBC-young boost; 2003-13 (Other Grant/Funding Number: Commissie Klinische Studies)
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Breast Cancer
Keywords: breast cancer; radiotherapy; microarrays
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): low dose boost (16 Gy)
  Interventions: Radiation: high dose boost; Procedure: boost
- 2 (Experimental): high boost (26 Gy)
  Interventions: Radiation: high dose boost; Procedure: boost

INTERVENTIONS:
Radiation: high dose boost — high dose boost
Procedure: boost — low dose versus high dose

SUMMARY:
hypothesis: 10 Gy additional boost to the tumor bed will yield an increase in local control at 10 years from 88% to 93%, with still acceptable cosmesis.

DETAILED DESCRIPTION:
Title of the study:

Radiation dose intensity study in breast cancer in young women: a randomized phase III trial of additional dose to the tumor bed.

Background and aim of the study:

Several studies showed that breast conserving therapy (BCT) yields similar survival rates as mastectomy. BCT consists of lumpectomy followed by whole breast radiotherapy (WBRT). Three studies showed that an additional dose to the tumor bed, after 50 Gy WBRT, reduces the local recurrence rate (LRR). The largest of these 3 studies was a recent EORTC trial, which also showed that young age was an independent risk factor for LR after BCT.

In patients < 51 years of age, the LR rate was reduced with 50% after a 66 Gy dose to the tumor bed, compared to 50 Gy (5-year LRR 12% vs 5.9%, p < 0.02). However, the LRR in young women was still quite high (> 1% per year). Therefore the first aim of the study is to investigate whether an additional boost dose to the tumorbed (26 Gy) reduces the LRR further. Therefore, we will compare the effect of a low boost dose (16 Gy) with the effect of a high boost dose (26 Gy) on the LRR, but also on the cosmetic outcome.

The second, very important aim of this study is to investigate whether we can find genetic or protein profiles that correlate with LRR, lymph node metastases, distant metastases, survival, radiosensitivity, and age. For this purpose we will obtain frozen tumor material and blood samples of as many patients as possible.

Population, study design, intervention:

Patients younger than 51 years of age, with stage T1-2N01-2aM0 breast cancer, and where the tumor can be locally excised with acceptable cosmetic result, will be randomized between a 16 Gy boost dose to the tumorbed and a 26 Gy boost dose to the tumor bed, after 50 Gy WBRT. Patients will be stratified based on age, tumor size, lymph node metastases, estrogen receptor status, interstitial or external boost irradiation, and institution. In principle frozen tumor samples and blood samples will be stored of each patient.

Endpoints and statistics:

The primary endpoint is LRR are 10 years. The secondary endpoint is cosmetic result, which will be quantified using digitized color photographs. In addition, patients will be asked to give their opinion about the cosmetic result using standardized questionnaires.

To find an increase in the local control rate of 88% to 93% at 10 year, with a power of 80% and a significance level of 5%, 580 patients will be included in each treatment arm.

Side studies:

An extremely important aspect of this trial is to obtain fresh tumor material and blood samples. These will be used to determine genetic and protein profiles aimed at finding subgroups based on these profiles, which may take more or less advantage of the additional radiation treatment.

ELIGIBILITY:
Inclusion criteria:

* Age 50 years or younger.
* Histological diagnosis of invasive mammary cancer including all subtypes of invasive adenocarcinoma.
* Tumor location and extension imaged prior to surgery using at least mammography and ultrasound.
* Unicentric tumors and multifocal tumors removed using a wide local excision; microscopic radical resection (focally involved margins allowed, defined as:

any DCIS or invasive carcinoma in 3 or fewer low-power fields (using a x 4 objective and a x 10 ocular lens, which has a diameter of 5 mm per low-power microscopic fields).

* Sentinel lymph node biopsy and/or axillary lymph node dissection has been performed.
* Breast cancer stage: pT1-2pN0-2a M0.
* No treatment is allowed prior to surgery (no neoadjuvant chemotherapy, no neoadjuvant hormonal therapy, no pre-operative radiotherapy).
* In cases where no adjuvant chemotherapy is given, wide local excision has been performed < 10 weeks before the start of radiotherapy.
* In cases where adjuvant chemotherapy is given immediately after surgery, wide local excision has been performed < 6 months before the start of radiotherapy, and chemotherapy should be completed < 6 weeks before the start of radiotherapy.
* In cases where hormonal treatment is planned, this is given after completion of the radiotherapy.
* No previous history or synchronous malignant tumor in the other breast, previous history of malignant disease, except adequately treated carcinoma in situ of the cervix or basal cell carcinoma of the skin.
* ECOG performance scale 2 or less.

Exclusion criteria:

* Residual microcalcifications on mammogram.
* All histological types of malignancies other than invasive adenocarcinoma.
* In situ carcinoma of the breast, without invasive tumor.
* Concurrent pregnancy.
* Multicentric tumors, and multifocal. tumors excised using multiple excisions * Invasive breast cancer in both breasts.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2400 (Estimated)
Dates: Start 2004-07; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Local control at 10 yr | at every follow up visit (< 2 months after last radiation treatment and thereafter yearly

SECONDARY OUTCOMES:
Cosmetic outcome | prior to radiotherapy, 1 year after radiotherapy and thereafter every 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Liesbeth Boersma, MD, Study Chair — MAASTRO Clinic, Heerlen
Locations (18):
- France (17):
  - Hôpital J-Minjoz, Besançon
  - Institut Bergonié, Bordeaux
  - CHU Henri Mondor, Créteil
  - Centre Oscar Lambret, Lille
  - Institut Paoli Calmettes, Marseille
  - Centre Val d'Aurelle, Montpellier
  - Centre Antoine Lacassagne, Nice
  - Institut Curie, Paris
  - Hôpital Saint Louis, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Centre Eugène Marquis, Rennes
  - Centre Henri Becquerel, Rouen
  - Centre René Huguenin, Saint-Cloud
  - Centre René Gauducheau, Saint-Herblain
  - Centre Paul Strauss, Strasbourg
  - CHU de Tours, Tours
  - Institut Gustave Roussy, Villejuif
- The Netherlands Cancer Institute, Amsterdam, Netherlands